CLINICAL TRIAL: NCT06308588
Title: Phase I/II Study of the Combination of Blinatumomab and Asciminib in Patients With Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0054; NCI-2024-02121 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Philadelphia Chromosome-Positive; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blinatumomab + Asciminib (Experimental): Participants found to be eligible to take part in this study will receive 5 cycles of blinatumomab and asciminib, followed by asciminib alone for as long as it benefits the participant.
  Participants will receive blinatumomab as a continuous (non-stop) infusion on Days 4-31 of Cycle 1 and on Days 1-28 of Cycles 2-5.
  Participants will take asciminib by mouth 2 times every day during this study.
  Interventions: Drug: Blinatumomab; Drug: Asciminib

INTERVENTIONS:
Drug: Blinatumomab — Given by Infusion
Drug: Asciminib — Given by PO
  Other Names: ABL001

SUMMARY:
To learn if the combination of blinatumomab and asciminib can help to control Ph+ ALL.

DETAILED DESCRIPTION:
Primary Objectives

* Phase I: To determine the minimum safe and biologically effective dose of asciminib in combination with blinatumomab
* Phase II: To evaluate the rate of NGS measurable residual disease (MRD) negativity using the clonoSEQ® assay in cohort 1 (newly diagnosed Ph-positive ALL) and the overall response (CR+CRi) rate in cohort 2 (relapsed/refractory disease).

Secondary Objectives

* To evaluate other clinical efficacy endpoints (complete molecular response [CMR] rate, CR rate, relapse-free survival and overall survival)
* To determine the safety of the combination regimen

Exploratory Objectives

* To characterize the role of ABL1 kinase domain mutations on treatment failure and relapse
* To assess concordance/discordance between MRD assessed by PCR for BCR::ABL1 and next-generation sequencing MRD
* To determine the effect of the combination regimen on immune cell subsets

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of one of the following:

   a) Participants ≥18 years of age with previously untreated or minimally pretreated Ph-positive ALL who are not suitable candidates for intensive chemotherapy. Participants who have received no more than one or two courses of chemotherapy with or without other TKIs are considered minimally pretreated and still eligible if they have persistently detectable MRD.

   i. If they are in morphologic remission at enrollment, they are evaluable only MRD responses, RFS and OS b) Participants ≥ 12 years of age with relapsed/refractory Ph-positive ALL or with previously treated lymphoid blast phase CML
2. Performance status ≤2 (ECOG Scale) if age ≥18 years or Lansky ≥50 if age <18 years
3. Weight ≥40kg
4. Adequate liver function as defined by the following criteria (unless the increased values are judged to be leukemia disease related):

   1. Total serum bilirubin ≤ 2 x upper limit of normal (ULN), unless due to Gilbert's syndrome
   2. Alanine aminotransferase (ALT) ≤ 3 x ULN, OR
   3. Aspartate aminotransferase (AST) ≤ 3 x ULN
5. Adequate renal function defined as:

   a) Creatinine clearance ≥30 mL/min
6. Adequate pancreatic function as defined by the following criteria:

   a) Serum lipase and amylase < 1.5 x ULN
7. Adequate cardiac function as assessed clinically by history and physical examination.
8. For females of childbearing potential, a negative urine pregnancy test must be documented
9. Willingness to use adequate contraception prior to study entry, for the duration of study participation, and for 4 months after completion of study participation. For women of child-bearing potential, adequate methods of contraception include: complete abstinence, hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), intrauterine device (IUD), tubal Ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide
10. Ability to understand and the willingness to sign a written informed consent document.
11. Signed informed consent

Exclusion Criteria:

1. Active serious infection not controlled by oral or intravenous antibiotics.
2. Active secondary malignancy other than skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year.
3. Active Grade III-V cardiac failure as defined by the New York Heart Association Criteria.
4. Prolonged QTc interval on pre-entry electrocardiogram (> 470 msec) unless corrected after electrolyte replacement or approved by cardiologist
5. History or presence of clinically relevant CNS pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis. (Participants with active CNS leukemia will NOT be excluded)
6. Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator. Cytarabine 2 g/m2 (or alternative) for cytoreduction is permitted.
7. Pregnant and lactating women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Short, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT06308588/ICF_000.pdf